CLINICAL TRIAL: NCT05325463
Title: Safety and Efficacy of Ultrasound-guided Lung Recruitment Maneuvers for Prevention of Postoperative Atelectasis After Surgical Correction of Idiopathic Adolescent Scoliosis. A Prospective Randomized Study
Brief Title: Lung Recruitment Maneuvers for Postoperative Atelectasis Prevention After Idiopathic Adolescents' Scoliosis Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Atelectasis in scoliosis
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Atelectasis; Lung Recruitment; Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional (Experimental)
  Interventions: Procedure: conventional lung recruitment
- ultrasound- guided (Active Comparator)
  Interventions: Procedure: ultrasound- guided lung recruitment

INTERVENTIONS:
Procedure: conventional lung recruitment — The recruitment maneuver will be performed by pressure controlled mode maintaining a steady airway pressure of 15 cmH2O, with 5 cmH2O increments in positive end-expiratory pressure (PEEP) until a peak pressure of 30 cmH2O will be achieved. Each PEEP level will be maintained for 5 sec. The peak airway pressure will be maintained for 10 sec or five breaths and subsequently reduced, followed by maintenance with the previous ventilator settings.
  Arms: conventional
Procedure: ultrasound- guided lung recruitment — The recruitment maneuver will be performed under ultrasound guidance until no collapsed lung area was visible. The strategy to increase the airway pressure will be the same as that for the conventional maneuver, although the maximal pressure limit was 40 cmH2O.
  Arms: ultrasound- guided

SUMMARY:
The investigators hypothesized that an ultrasound-guided lung recruitment maneuvers would be more effective in preventing postoperative atelectasis than conventional alveolar recruitment after surgical correction of idiopathic adolescent scoliosis.

DETAILED DESCRIPTION:
In anesthetized children, the incidence of lung collapse with episodes of hypoxemia is high. Diaphragm dysfunction induced by general anesthesia is one of the most important factors in the genesis of regional losses of lung aeration; the mass of the abdominal organs pushes the diaphragm cranially compressing the lungs in the most dependent areas. Such regional lung collapse may range from slight loss of aeration to complete atelectasis.

Scoliosis correction surgery for adolescent idiopathic scoliosis (AIS) is effective in preventing deterioration of lung function caused by disease progression, and improving lung volume over the long term. However, complications of the respiratory system and pulmonary dysfunction may occur in the immediate postoperative period. General anesthesia (GA) and positive pressure ventilation can cause decreased lung volumes, expiratory flow rates, and oxygenation after surgery as a result of positive pressure ventilation, partial recovery of respiratory muscle, pain, and immobilization.

Lung ultrasound has been gaining consensus as a noninvasive, radiation-free tool for diagnosing various pulmonary diseases in adult and pediatric patients. Evidence supporting lung ultrasound use is expanding beyond emergency and critical care settings to perioperative care.

It has been reported that lung ultrasound (LUS) at a patient's bedside immediately following surgery can be useful for diagnosing respiratory complications. LUS has proven to be a valuable bedside diagnostic tool for pneumothorax, with high sensitivity and specificity (78.6% and 98.4%, respectively), and a higher rate of detecting abnormalities such as lung alveolar consolidation and pleural effusion than bedside chest X-ray or physical examination. LUS has also been used to diagnose anesthesia-induced atelectasis in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective correction of AIS
* aged between 10 and 25 years old
* American society of anesthesiologists (ASA) class I & II
* both genders

Exclusion Criteria:

* Morbidly obese patients
* patients with previous thoracic surgery
* upper or lower airway infection within 2 weeks before the surgery
* abnormal preoperative chest x-ray findings including atelectasis, pneumothorax, pleural effusion or pneumonia

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
the incidence of atelectasis | postoperative first 2 hours
  the incidence of postoperative atelectasis in post-anaesthesia care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Tanta university, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No